CLINICAL TRIAL: NCT02788864
Title: A Randomized, Placebo-controlled, Double-blind Trial Using Dihydroartemisinine+Piperaquine (DP) to Protect Forest Workers From Malaria in Bu Gia Map National Park
Brief Title: Prevention of Malaria With Dihydroartemisinine + Piperaquine for Forest Rangers
Acronym: PREMAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oxford University Clinical Research Unit, Vietnam (Other)
Collaborators: Binh Phuoc Malaria Control Centre (Unknown); Bu Gia Map National Park, Binh Phuoc Province, Vietnam (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17MA
Record Dates: First submitted 2016-05-27; First posted 2016-06-02 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Malaria
Keywords: Forest ranger; P.falciparum; P.vivax; Dihydroartemisinine-piperaquine (DP); Primaquine
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arterakine (Active Comparator): Active drug: Arterakine (DHA/piperaquine) one tablet contains 40 mg of dihydroartemisinin and 320 mg piperaquine. Weight based regimen: 7 mg/kg dihydroartemisinin; 55 mg/kg piperaquine phosphate) for 3 days prior to forest visit (day -2, -1 and day 0 prior forest visit)
  Interventions: Drug: Arterakine (DHA/piperaquine)
- Placebo (Placebo Comparator): Placebo (visually matched to Arterakine for 3 days prior to forest visit (day -2, -1 and day 0 prior forest visit)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Arterakine (DHA/piperaquine) — Stage 1: Parasite Clearance
  * Arterakine (DHA/piperaquine), one tablet contains 40 mg of dihydroartemisinine and 320 mg piperaquine. Weight based regimen: 7 mg/kg dihydroartemisinine; 55 mg/kg piperaquine phosphate) for 3 days
  * Primaquine (One tablet contains 13.2mg primaquine disphosphate/7.5mg base. Weight based regimen: 0.25mg base/kg) for 14 days
  Stage 2: Forest trip
  • Arterakine (DHA/piperaquine), one tablet contains 40 mg of dihydroartemisinine and 320 mg piperaquine. Weight based regimen: 7 mg/kg dihydroartemisinine; 55 mg/kg piperaquine phosphate) for 3 days prior to forest visit (day -2, -1 and day 0 prior forest visit)
  Arms: Arterakine
Drug: Placebo — Stage 1: Parasite Clearance
  * Arterakine (DHA/piperaquine), one tablet contains 40 mg of dihydroartemisinine and 320 mg piperaquine. Weight based regimen: 7 mg/kg dihydroartemisinine; 55 mg/kg piperaquine phosphate) for 3 days
  * Primaquine (One tablet contains 13.2mg primaquine disphosphate/7.5mg base. Weight based regimen: 0.25mg base/kg) for 14 days
  Stage 2: Forest trip
  • Placebo (visually matched to Arterakine (DHA/piperaquine) for 3 days prior to forest visit (day -2, -1 and day 0 prior forest visit)
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess if the antimalarial drugs Dihydroartemisinine + Piperaquine (DP) are effective in preventing malaria infection for forest ranger

DETAILED DESCRIPTION:
To assess the protective effect of 3-day DP regimen for forest rangers working for long-term in forest where malaria transmission is intense, all eligible forest rangers will be treated with a full course of DP + primaquine to eradicate all parasites which may survive in their blood while staying in non- malaria transmission areas.

Just before returning back to the forest participants will be randomized to receive either Arterakine (dihydroartemisinine (DHA)/piperaquine) (intervention arm) or placebo (control arm). Participants will be assessed for parasitemia before and after the forest trip with high volume, ultrasensitive, PCR (HVUqPCR). The minimum time span between two forest trips should be 20 days so participants could complete the 14 day primaquine course and the Arterakine (dihydroartemisinine (DHA)/piperaquine).

There is no limit in the duration between trips. Participants are tested for P.falciparum, P.vivax infection before they return to the forest.

Each participant will be visited 2 weeks or later after returning home from the forest and examined. The rationale for the added two weeks is to detect blood stages of infections, which may have been inoculated towards the end of the forest visit.

If found to be sick, the patient will be treated according to government treatment guidelines. A 4ml venous blood sample will be obtained for Hb and HVUSqPCR.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Male, over or equal to18 years of age
3. Able and willing to comply with the study requirements and follow-up

Exclusion Criteria:

1. Inability to tolerate oral treatment
2. Previous episode of haemolysis or severe haemoglobinuria following primaquine
3. Glucose-6-phosphate dehydrogenase (G6PD) deficient with Hb < 9 g/dL *
4. Known hypersensitivity or allergy to any study drugs * If the participant with G6PD deficient gets malaria, primaquine would be used as recommended by World Health Organization (WHO) (once a week for 8 weeks) in combination with 3 days of chloroquine.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
the proportion of study subjects with any malaria parasitaemia (P.falciparum, mixed parasitaemia of P.falciparum and P.vivax) and the incidence rate of symptomatic malaria | at 2 weeks after coming back from the forest
  The primary endpoints are the proportion of study subjects with any malaria parasitaemia (P.falciparum, mixed parasitaemia of P.falciparum and P.vivax) at 2 weeks after coming back from the forest assessed by high volume, ultrasensitive PCR (HVUSqPCR) and the incidence rate of symptomatic malaria (P.falciparum, mixed P.falciparum + P.vivax) during the two week follow-up period as assessed by the study doctor.

SECONDARY OUTCOMES:
The proportion of different anopheles species amongst all captured mosquito anopheles | 1 month
  The proportion of different anopheles species amongst all captured mosquito anopheles as identified by morphology
The proportion of sporozoite-carrying mosquitoes (any parasite, P.falciparum, mixed P.falciparum and P.vivax) | 6 months
  The proportion of sporozoite-carrying mosquitoes (any parasite, P.falciparum, mixed P.falciparum and P.vivax) as assessed by PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Hung Son Do, Dr, Principal Investigator — Oxford University Clinical Research Unit
Locations (1):
- Bu Gia Map Commune Health Station, Bình Phước, Binh Phuoc, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data will be made available to researcher and public as a supporting material via open access journal and/or upon request by qualified research groups.

REFERENCES:
- [Background] Thanh PV, Van Hong N, Van Van N, Van Malderen C, Obsomer V, Rosanas-Urgell A, Grietens KP, Xa NX, Bancone G, Chowwiwat N, Duong TT, D'Alessandro U, Speybroeck N, Erhart A. Epidemiology of forest malaria in Central Vietnam: the hidden parasite reservoir. Malar J. 2015 Feb 19;14:86. doi: 10.1186/s12936-015-0601-y. PMID 25880664
- [Background] Parker DM, Carrara VI, Pukrittayakamee S, McGready R, Nosten FH. Malaria ecology along the Thailand-Myanmar border. Malar J. 2015 Oct 5;14:388. doi: 10.1186/s12936-015-0921-y. PMID 26437860
- [Background] Abe T, Honda S, Nakazawa S, Tuong TD, Thieu NQ, Hung le X, Thuan le K, Moji K, Takagi M, Yamamoto T. Risk factors for malaria infection among ethnic minorities in Binh Phuoc, Vietnam. Southeast Asian J Trop Med Public Health. 2009 Jan;40(1):18-29. PMID 19323029
- [Background] Sanh NH, Van Dung N, Thanh NX, Trung TN, Van Co T, Cooper RD. Forest malaria in central Vietnam. Am J Trop Med Hyg. 2008 Nov;79(5):652-4. PMID 18981498
- [Background] Erhart A, Ngo DT, Phan VK, Ta TT, Van Overmeir C, Speybroeck N, Obsomer V, Le XH, Le KT, Coosemans M, D'alessandro U. Epidemiology of forest malaria in central Vietnam: a large scale cross-sectional survey. Malar J. 2005 Dec 8;4:58. doi: 10.1186/1475-2875-4-58. PMID 16336671
- [Background] Erhart A, Thang ND, Hung NQ, Toi le V, Hung le X, Tuy TQ, Cong le D, Speybroeck N, Coosemans M, D'Alessandro U. Forest malaria in Vietnam: a challenge for control. Am J Trop Med Hyg. 2004 Feb;70(2):110-8. PMID 14993619
- [Background] Imwong M, Nguyen TN, Tripura R, Peto TJ, Lee SJ, Lwin KM, Suangkanarat P, Jeeyapant A, Vihokhern B, Wongsaen K, Van Hue D, Dong le T, Nguyen TU, Lubell Y, von Seidlein L, Dhorda M, Promnarate C, Snounou G, Malleret B, Renia L, Keereecharoen L, Singhasivanon P, Sirithiranont P, Chalk J, Nguon C, Hien TT, Day N, White NJ, Dondorp A, Nosten F. The epidemiology of subclinical malaria infections in South-East Asia: findings from cross-sectional surveys in Thailand-Myanmar border areas, Cambodia, and Vietnam. Malar J. 2015 Sep 30;14:381. doi: 10.1186/s12936-015-0906-x. PMID 26424000
- [Background] Imwong M, Hanchana S, Malleret B, Renia L, Day NP, Dondorp A, Nosten F, Snounou G, White NJ. High-throughput ultrasensitive molecular techniques for quantifying low-density malaria parasitemias. J Clin Microbiol. 2014 Sep;52(9):3303-9. doi: 10.1128/JCM.01057-14. Epub 2014 Jul 2. PMID 24989601
- [Derived] Son DH, Thuy-Nhien N, von Seidlein L, Le Phuc-Nhi T, Phu NT, Tuyen NTK, Tran NH, Van Dung N, Van Quan B, Day NPJ, Dondorp AM, White NJ, Thwaites GE, Hien TT. The prevalence, incidence and prevention of Plasmodium falciparum infections in forest rangers in Bu Gia Map National Park, Binh Phuoc province, Vietnam: a pilot study. Malar J. 2017 Nov 6;16(1):444. doi: 10.1186/s12936-017-2091-6. PMID 29110709